CLINICAL TRIAL: NCT01427725
Title: Special Investigation of LipaCreon on Long-term Use in Patients With Pancreatic Exocrine Insufficiency Due to Chronic Pancreatitis, Pancreatectomy and Other Conditions Except Cystic Fibrosis
Brief Title: Special Investigation of LipaCreon on Long-term Use in Patients With Pancreatic Exocrine Insufficiency
Status: Completed | Type: Observational
Sponsor: Mylan Inc. (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Other Study IDs: P12-894
Record Dates: First submitted 2011-08-31; First posted 2011-09-02 (Estimated); Results first posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-03

CONDITIONS: Exocrine Pancreatic Insufficiency; Pancreatic Diseases; Digestive System Diseases
Keywords: Digestive System Diseases; Therapeutic Uses; Pancreatectomy; Gastrointestinal Agents; Pancreatic Diseases; Pancrelipase; Exocrine Pancreatic Insufficiency
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Pancreatic Diseases; Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lipacreon: In general, pancrelipase 600 mg/dose was orally administered immediately after a meal, 3 times a day.
  Also, the dose was adjusted appropriately according to the patient's condition.
  Interventions: Drug: Lipacreon

INTERVENTIONS:
Drug: Lipacreon — This study was an observational study and no intervention was specified

SUMMARY:
This study aims at collecting the information related to the safety and effectiveness in the pancreatic exocrine insufficiency patients receiving the treatment with LipaCreon for a long term in order to evaluate the effective and safe use of LipaCreon.

DETAILED DESCRIPTION:
Criteria for evaluation:

1. Adverse events
2. Nutritional endpoints

   * BMI (height [only prior to the start of Lipacreon treatment] and weight)
   * Serum total protein
   * Albumin
   * Total cholesterol
   * Triglycerides
   * Haemoglobin
3. Symptoms related to exocrine pancreatic insufficiency

   * Steatorrhoea
   * Frequency of bowel movements
   * Diarrhoea
   * Foul stool odour
   * Decreased appetite
   * Abdominal distension
4. Patient's quality of life (QOL)
5. Degree of general improvement

ELIGIBILITY:
Inclusion Criteria

* Patients who receive LipaCreon for the replacement of pancreatic digestive enzymes in pancreatic exocrine insufficiency

Exclusion Criteria

* Patients with a history of hypersensitivity to the ingredient of LipaCreon.
* Patients with a history of hypersensitivity to porcine protein.

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who receive LipaCreon for the replacement of pancreatic digestive enzymes in pancreatic exocrine insufficiency
Sampling Method: Non-Probability Sample
Enrollment: 579 (Actual)
Dates: Start 2011-09; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Kato, MD.,Ph.D., Study Director — Abbott Japan Co.,Ltd
Locations (189):
- Japan (189):
  - Research facility ID ORG-000247, Aichi
  - Research facility ID ORG-000216, Aichi
  - Research facility ID ORG-000214, Aichi
  - Research facility ID ORG-000215, Aichi
  - Research facility ORG-000096, Aichi
  - Research facility ORG-000086, Aichi
  - Research facility ORG-000120, Aichi
  - Research facility ORG-000119, Aichi
  - Research facility ID ORG-000208, Aichi
  - Site reference ID/Investigator # 75775, Aichi
  - Research facility ID ORG-000256, Aichi
  - Site Reference ID/Investigator# 68371, Akita
  - Site Reference ID/Investigator# 71098, Akita
  - Research facility ORG-000222, Akita
  - Research facility ORG-000129, Aomori
  - Research facility ORG-000133, Aomori
  - Site Reference ID/Investigator# 68378, Chiba
  - Site Reference ID/Investigator# 75790, Chiba
  - Research facility ORG-000162, Chiba
  - site REference ID/Investigator# 75798, Chiba
  - Research facility ID ORG-000246, Chiba
  - Site reference ID/Investigator# 88676, Chiba
  - Research facility ORG-000118, Chiba
  - Research facility ID ORG-000251, Ehime
  - Research facility ID ORG-000232, Ehime
  - Research facility ORG-000233, Ehime
  - Research facility ORG-000130, Ehime
  - Research facility ID ORG-000271, Fukui
  - Site reference ID/Investigator # 88674, Fukui
  - Research facility ORG-000094, Fukuoka
  - Research facility ID ORG-000269, Fukuoka
  - Investigator ID 117496, Fukuoka
  - Research facility ID ORG-000229, Fukuoka
  - Research facility ORG-000088, Fukuoka
  - Research facility ORG-000098, Fukuoka
  - Research facility ORG-000104, Fukuoka
  - Research facility ORG-000091, Fukuoka
  - Research facility ORG-000165, Fukuoka
  - Research facility ID ORG-000262, Fukuoka
  - Research facility ORG-000114, Fukuoka
  - Site Reference ID/Investigator# 84554, Fukushima
  - Research facility ID ORG-000207, Fukushima
  - Research facility ORG-000136, Fukushima
  - Research facility ID ORG-000177, Fukushima
  - Research facility ID ORG-000238, Gifu
  - Site reference ID/Investigator# 91833, Gifu
  - Research facility ORG-000139, Gunma
  - Research facility ID ORG-000272, Gunma
  - Site reference ID/Investigator # 84557, Gunma
  - Research facility ORG-000156, Hiroshima
  - Research facility ID ORG-000241, Hiroshima
  - Research facility ID ORG-000203, Hiroshima
  - Site reference ID/Investigator # 91835, Hiroshima
  - Site Reference ID/Investigator# 88698, Hiroshima
  - Site Reference ID/Investigator# 84515, Hiroshima
  - Research facility ORG-000155, Hiroshima
  - Research facility ID ORG-000213, Hokkaido
  - Research facility ORG-000097, Hokkaido
  - Research facility ID ORG-000220, Hokkaido
  - Research facility ID/Investigator # ORG-000221 / 86896, Hokkaido
  - Site Reference ID/Investigator# 84535, Hokkaido
  - Research facility ID ORG-000250, Hokkaido
  - Site Reference ID# 84573, Hokkaido
  - Research facility ID ORG-000223, Hokkaido
  - Research facility ID ORG-000201, Hokkaido
  - Research facility ID ORG-000211, Hokkaido
  - Site reference ID/Investigator# 84575, Hokkaido
  - Research facility ORG-000140, Hokkaido
  - Research facility ORG-000142, Hyōgo
  - Research facility ID ORG-000225, Hyōgo
  - Research facility ORG-000159, Hyōgo
  - Research facility ORG-000160, Hyōgo
  - Research facility ORG-000163, Hyōgo
  - Site Reference ID/Investigator# 73816, Hyōgo
  - Research facility ORG-000152, Hyōgo
  - Site Reference ID/Investigator# 75804, Ibaraki
  - Research facility ID ORG-000249, Ibaraki
  - Research facility ID ORG-000181, Ibaraki
  - Investigator ID 117498, Ishikawa
  - Research facility ID ORG-000260, Kagawa
  - Research facility ORG-000107, Kagoshima
  - Site reference ID/Investigator# 91860, Kagoshima
  - Research facility ID ORG-000244, Kagoshima
  - Research facility ID ORG-000273, Kagoshima
  - Research facility ID ORG-000212, Kanagawa
  - Research facility ID ORG-000167, Kanagawa
  - Research facility ID ORG-000202, Kanagawa
  - Research faciliity ORG-000099, Kanagawa
  - Research facility ID ORG-000191, Kanagawa
  - Research facility ID ORG-000182, Kanagawa
  - Research facility ID ORG-000255, Kanagawa
  - Research facility ID ORG-000254, Kanagawa
  - Site reference ID/Investigator # 75802, Kanagawa
  - Research facility ORG-000154, Kochi
  - Research facility ID ORG-000166, Kochi
  - Research facility ORG-000113, Kumamoto
  - Site reference ID/Investigator # 75789, Kyoto
  - Research facility ORG-000150, Kyoto
  - Research facility ID ORG-000176, Kyoto
  - Research facility ORG-000153, Kyoto
  - Research faclity ORG-000112, Kyoto
  - Research facility ID ORG-000180, Kyoto
  - Research facility ID ORG-000196, Kyoto
  - Investigator ID 117503, Kyoto
  - Research facility ID ORG-000194, Kyoto
  - Research facility ID ORG-000237, Mie
  - Research facility ORG-000105, Mie
  - Research facility ORG-000147, Miyagi
  - Research facility ORG-000092, Miyagi
  - Research facility ORG-000093, Miyagi
  - Site reference ID/Investigator # 84561, Miyagi
  - Site Reference ID/Investigator# 84560, Miyagi
  - Investigator ID 117508, Miyazaki
  - Investigator ID 117507, Miyazaki
  - Site reference ID/Investigator# 96736, Nagano
  - Research facility ORG-000171, Nagano
  - Research facility ID ORG-000290, Nagano
  - Research facility ORG-000109, Nagano
  - Research facility ORG-000115, Nagano
  - Research facility ORG-000137, Nagasaki
  - Site reference ID/Investigator # 71102, Nara
  - Research facility ID ORG-000265, Nara
  - Research facility ORG-000100, Niigata
  - Research facility ORG-000102, Niigata
  - Research facility ORG-000267, Niigata
  - Research facility ID ORG-000193, Niigata
  - Site Reference ID/Investigator# 63982, Numakunai
  - Site reference ID/Investigator # 91836, Okayama
  - Research facility ORG-000268, Okayama
  - Research facility ID ORG-000231, Okayama
  - Site reference ID/Investigator # 91856, Okinawa
  - Site Reference ID/Investigator# 86894, Osaka
  - Research facility ORG-000117, Osaka
  - Research facility ORG-000095, Osaka
  - Research facility ID ORG-000183, Osaka
  - Research facility ORG-000089, Osaka
  - Research facility ORG-000090, Osaka
  - Research facility ORG-000106, Ōita
  - Investigator ID 117497, Ōita
  - Research facility ID ORG-000204, Saga
  - Research facility ORG-000157, Saitama
  - Research facility ORG-000143, Saitama
  - Research facility ID ORG-000189, Saitama
  - Research facility ORG-000135, Saitama
  - Research facility ID ORG-000190, Saitama
  - Research facility ID ORG-000173, Saitama
  - Research facility ID ORG-000199, Saitama
  - Site Reference ID/Investigator# 86895, Saitama
  - Research facility ORG-000172, Saitama
  - Site reference ID/Investigator# 96739, Saitama
  - Research facility ORG-000116, Shiga
  - Research facility ID ORG-000178, Shimane
  - Research facility ID ORG-000253, Shizuoka
  - Research facility ID ORG-000252, Shizuoka
  - Site Reference ID/Investigator# 91834, Shizuoka
  - Site reference ID/Investigator# 84576, Shizuoka
  - Research facility ID ORG-000239, Shizuoka
  - Research facility ORG-000126, Tochigi
  - Research facility ORG-000108, Tochigi
  - Research facility ORG-000146, Tokyo
  - Research facility ORG-000124, Tokyo
  - Research facility ORG-000132, Tokyo
  - Research facility ORG-000121, Tokyo
  - Research facility ORG-000164, Tokyo
  - Site Reference ID/Investigator# 84578, Tokyo
  - Investigator ID 117499, Tokyo
  - Research facility ORG-000110, Tokyo
  - Research facility ORG-000101, Tokyo
  - Site Reference ID/Investigator# 73824, Tokyo
  - Investigator ID 117504, Tokyo
  - Investigator ID 117505, Tokyo
  - Research facility ID ORG-000179, Tokyo
  - Research facility ORG-000138, Tokyo
  - Research facility ID ORG-000195, Tokyo
  - Research facility ORG-000161, Tokyo
  - Research facility ORG-000123, Tokyo
  - Site Reference ID/Investigator# 75777, Tokyo
  - Research facility ID ORG-000227, Tokyo
  - Research facility ORG-000158, Tokyo
  - Research facility ORG-000103, Tokyo
  - Investigator ID 117501, Tokyo
  - Research facility ORG-000151, Tokyo
  - Site reference ID/Investigator # 86913, Tottori
  - Research facility ID ORG-000243, Wakayama
  - Research facility ORG-000122, Yamagata
  - Research facility ID ORG-000263, Yamaguchi
  - Research facility ORG-000128, Yamaguchi
  - Research facility ID ORG-000266, Yamaguchi
  - Research facility ORG-000127, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From August 30, 2011 to July 31, 2014, 579 patients were registered at 144 departments of 136 facilities (patient registration period: August 30, 2011 to July 31, 2014) and the survey forms of 562 patients were collected from 140 departments of 132 facilities.
Pre-assignment Details: For this survey, the contract for the conduct of the survey was concluded with 190 departments of 181 facilities during the period from August 30, 2011 to July 31, 2014.
Groups:
- LipaCreon: those with an exposure
Period: Overall Study
Arm/Group | LipaCreon
Started | 579
Collected CRFs | 562 (Not collected Case Report Forms (CRFs) of 17 patients.)
Safety Analysis Set | 553 (Analysis of safety data. 9 patients dropped out, could not confirm existence of Adverse Events.)
Completed | 378 (Among the patients in the safety analysis set, 175 patients discontinued the survey.)
Not Completed | 201
Not completed — Lost to Follow-up | 17
Not completed — Protocol Violation | 1
Not completed — Drug not administered | 1
Not completed — Failure to visit | 7
Not completed — Adverse Event | 46
Not completed — Failure to visit after administration | 40
Not completed — Patient's rejection | 27
Not completed — Transfer to a different hospital | 17
Not completed — Lack of Efficacy | 8
Not completed — Death | 7
Not completed — Symptom improvement | 6
Not completed — AE and Patient's rejection | 5
Not completed — Physician Decision | 5
Not completed — Exacerbation of underlying disease | 5
Not completed — Oral feeding difficulty | 5
Not completed — Lack of Efficacy and Patient's rejection | 1
Not completed — Forgetting prescription | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: 553 are effctive number for safety analysis
Arm/Group | LipaCreon
Number analyzed (Participants) | 553
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 243
  >=65 years | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210
  Male | 343
Region of Enrollment [Number; unit: participants]
  Japan | 553

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Drug Reaction
Description: An adverse event (AE) was defined as any unfavourable or unintended disease, or symptom or sign of such a disease, or abnormal laboratory finding that occurred in a patient who received Lipacreon, whether or not considered related to the medicinal product. Also, an AE for which the relationship with Lipacreon could not be ruled out was regarded as an adverse drug reaction (ADR).
  1. Related : There is a temporal relationship between the use of the medicinal product and the onset of an AE, or a relapse with readministration,where other factors are less likely to be involved.
  2. Relationship cannot be ruled out : There are other potential factors although there is a temporal relationship between the use of the medicinal product and the onset of an AE
Time Frame: At week 52
Measure: Number; unit: participants
Arm/Group | LipaCreon
Number analyzed (Participants) | 553
participants | 36

2. Secondary Outcome: Degree of General Improvement
Description: It was assessed at 24 weeks after the start of Lipacreon treatment and at the end of the observation period, using the following 4 grades:
  Improved, unchanged, exacerbated, unassessable
Time Frame: At week 24
Population: Among patients in the safety analysis set, 547 patients were included in the efficacy analysis set, excluding 6 patients who were excluded from the efficacy analysis set (Reasons: Unassessable: 5 patients; and off-label use: 1 patient). Among patients in the 547 patients, the patients for which data were obtained at each time frame were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Lipacreon: In general, pancrelipase 600 mg/dose was orally administered immediately after a meal, 3 times a day.
  Also, the dose was adjusted appropriately according to the patient's condition.
  Lipacreon: This study was an observational study and no intervention was specified
Arm/Group | Lipacreon
Number analyzed (Participants) | 404
Participants
  Improved | 299
  Unchanged | 87
  Exacerbated | 3
  Unassessable | 15

3. Secondary Outcome: Degree of General Improvement
Description: as for outcome 2
Time Frame: At week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Lipacreon
Number analyzed (Participants) | 314
Participants
  Improved | 240
  Unchanged | 62
  Exacerbated | 1
  Unassessable | 11

4. Secondary Outcome: Nutritional Endpoints - BMI
Description: The following nutritional endpoints were measured prior to the start of Lipacreon treatment, 4, 8 and 24 weeks after the start of treatment, and at the end of the observation period.
  * BMI (height [only prior to the start of Lipacreon treatment] and weight)
  * Serum total protein
  * Albumin
  * Total cholesterol
  * Triglycerides
  * Haemoglobin
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, and 52 weeks
Population: Among patients in the safety analysis set, 547 patients were included in the efficacy analysis set, excluding 6 patients who were excluded from the efficacy analysis set (Reasons: Unassessable: 5 patients; and off-label use: 1 patient). Among patients in the 547 patients, the patients for which data were obtained at each time frame were analyzed (Baseline:407 patients, 4 weeks:239 patients, 8 weeks:241 patients, 24 weeks:256 patients, 52weeks: 195 patients).
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
kg/m2
  Baseline: number analyzed (Participants) | 407
  Baseline | 20.452 (3.144)
  4 weeks: number analyzed (Participants) | 239
  4 weeks | 20.193 (2.933)
  8 weeks: number analyzed (Participants) | 241
  8 weeks | 20.229 (2.991)
  24 weeks: number analyzed (Participants) | 256
  24 weeks | 20.520 (2.847)
  52 weeks: number analyzed (Participants) | 195
  52 weeks | 20.720 (2.853)

5. Secondary Outcome: Nutritional Endpoints - Serum Total Protein
Description: as for outcome 4
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, and 52 weeks
Population: Among patients in the safety analysis set, 547 patients were included in the efficacy analysis set, excluding 6 patients who were excluded from the efficacy analysis set (Reasons: Unassessable: 5 patients; and off-label use: 1 patient). Among patients in the 547 patients, the patients for which data were obtained at each time frame were analyzed (Baseline:428 patients, 4 weeks:308 patients, 8 weeks:305 patients, 24 weeks:291 patients, 52weeks: 231 patients).
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
g/dL
  Baseline: number analyzed (Participants) | 428
  Baseline | 6.579 (0.798)
  4 weeks: number analyzed (Participants) | 308
  4 weeks | 6.955 (3.500)
  8 weeks: number analyzed (Participants) | 305
  8 weeks | 6.761 (0.654)
  24 weeks: number analyzed (Participants) | 291
  24 weeks | 6.901 (0.596)
  52 weeks: number analyzed (Participants) | 231
  52 weeks | 6.914 (0.637)

6. Secondary Outcome: Nutrition Endpoints - Albumin
Description: as for outcome 4
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, and 52 weeks
Population: Among patients in the safety analysis set, 547 patients were included in the efficacy analysis set, excluding 6 patients who were excluded from the efficacy analysis set (Reasons: Unassessable: 5 patients; and off-label use: 1 patient). Among patients in the 547 patients, the patients for which data were obtained at each time frame were analyzed (Baseline:429 patients, 4 weeks:319 patients, 8 weeks:316 patients, 24 weeks:309 patients, 52weeks: 235 patients).
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
g/dL
  Baseline: number analyzed (Participants) | 429
  Baseline | 3.688 (0.663)
  4 weeks: number analyzed (Participants) | 319
  4 weeks | 3.912 (2.164)
  8 weeks: number analyzed (Participants) | 316
  8 weeks | 3.843 (0.628)
  24 weeks: number analyzed (Participants) | 309
  24 weeks | 3.984 (0.509)
  52 weeks: number analyzed (Participants) | 235
  52 weeks | 3.959 (0.579)

7. Secondary Outcome: Nutrition Endpoints - Total Cholesterol
Description: as for outcome 4
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, and 52 weeks
Population: Among patients in the safety analysis set, 547 patients were included in the efficacy analysis set, excluding 6 patients who were excluded from the efficacy analysis set (Reasons: Unassessable: 5 patients; and off-label use: 1 patient). Among patients in the 547 patients, the patients for which data were obtained at each time frame were analyzed (Baseline:310 patients, 4 weeks:184 patients, 8 weeks:188 patients, 24 weeks:195 patients, 52weeks: 150 patients).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
mg/dL
  Baseline: number analyzed (Participants) | 310
  Baseline | 164.32 (47.63)
  4 weeks: number analyzed (Participants) | 184
  4 weeks | 169.40 (45.34)
  8 weeks: number analyzed (Participants) | 188
  8 weeks | 169.77 (45.99)
  24 weeks: number analyzed (Participants) | 195
  24 weeks | 168.88 (39.90)
  52 weeks: number analyzed (Participants) | 150
  52 weeks | 169.41 (38.27)

8. Secondary Outcome: Patient's Quality of Life - Physical Health (Summary)
Description: Baseline, 8 and 24 weeks after the start of treatment, and at the end of the observation period, the patient was asked to fill out the standard SF-8™ (1 month) to assess the patient's QOL, which was recorded in the survey form for this survey. SF-8™:The Medical Outcomes Study 8-Item Short-Form Health Survey (Japanese version). Items are as follows.
  Physical health (summary):PCS8, Mental health (summary):MCS8, General health:SF8GH, Physical functioning:SF8PF, Role physical:SF8RP, Body pain:SF8BP, Vitality:SF8VT, Social functioning:SF8SF, Mental health:SF8MH, Role emotional:SF8RE.
  PCS8 score is calculated by the following formula (All summed). PCS8 score = (0.23024×SF8GH)+(0.40672×SF8PF)+(0.38317×SF8RP)+(0.33295×SF8BP)+(0.07537×SF8VT)+(-0.01275×SF8SF)+(-0.30469×SF8MH)+(-0.14803×SF8RE)+0.67371
  The minimum value of PCS8 is 5.315, and the maximum value is 70.689. Higher scores mean a better outcome.
  The means ± SD was calculated by summing the values at each time point.
Time Frame: Baseline, 8 weeks, 24 weeks, and 52 weeks
Population: Among patients in the safety analysis set, 547 patients were included in the efficacy analysis set, excluding 6 patients who were excluded from the efficacy analysis set (Reasons: Unassessable: 5 patients; and off-label use: 1 patient). Among patients in the 547 patients, the patients for which data were obtained at each time frame were analyzed (Baseline:517 patients, 8 weeks:366 patients, 24 weeks:350 patients, 52weeks: 249 patients).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
score on a scale
  Baseline: number analyzed (Participants) | 517
  Baseline | 42.057 (9.590)
  8 weeks: number analyzed (Participants) | 366
  8 weeks | 46.086 (7.750)
  24 weeks: number analyzed (Participants) | 350
  24 weeks | 47.919 (7.414)
  52 weeks: number analyzed (Participants) | 249
  52 weeks | 48.985 (7.109)

9. Secondary Outcome: Symptoms Related to Exocrine Pancreatic Insufficiency - Steatorrhoea
Description: The following symptoms were assessed as those related to exocrine pancreatic insufficiency prior to the start of Lipacreon treatment, 4, 8 and 24 weeks after the start of treatment, and at the end of the observation period.
  * Steatorrhoea (Yes/No)
  * Frequency of bowel movements (times/day)
  * Diarrhoea (Yes/No)
  * Foul stool odour (Yes/No)
  * Decreased appetite (Yes/No)
  * Abdominal distension (Yes/No)
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, and 52 weeks
Population: Among patients in the safety analysis set, 547 patients were included in the efficacy analysis set, excluding 6 patients who were excluded from the efficacy analysis set (Reasons: Unassessable: 5 patients; and off-label use: 1 patient). Among patients in the 547 patients, the patients for which data were obtained at each time frame were analyzed (Baseline:470 patients, 4 weeks:363 patients, 8 weeks:355 patients, 24 weeks:347 patients, 52weeks: 276 patients).
Measure: Number; unit: participants
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
participants
  Baseline, Yes: number analyzed (Participants) | 470
  Baseline, Yes | 84
  Baseline, No: number analyzed (Participants) | 470
  Baseline, No | 386
  4 weeks, Yes: number analyzed (Participants) | 363
  4 weeks, Yes | 33
  4 weeks, No: number analyzed (Participants) | 363
  4 weeks, No | 330
  8 weeks, Yes: number analyzed (Participants) | 355
  8 weeks, Yes | 22
  8 weeks, No: number analyzed (Participants) | 355
  8 weeks, No | 333
  24 weeks, Yes: number analyzed (Participants) | 347
  24 weeks, Yes | 15
  24 weeks, No: number analyzed (Participants) | 347
  24 weeks, No | 332
  52 weeks, Yes: number analyzed (Participants) | 276
  52 weeks, Yes | 6
  52 weeks, No: number analyzed (Participants) | 276
  52 weeks, No | 270

10. Secondary Outcome: Nutrition Endpoints - Triglycerides
Description: as for outcome 4
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, and 52 weeks
Population: Among patients in the safety analysis set, 547 patients were included in the efficacy analysis set, excluding 6 patients who were excluded from the efficacy analysis set (Reasons: Unassessable: 5 patients; and off-label use: 1 patient). Among patients in the 547 patients, the patients for which data were obtained at each time frame were analyzed (Baseline:298 patients, 4 weeks:163 patients, 8 weeks:178 patients, 24 weeks:188 patients, 52weeks: 142 patients).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
mg/dL
  Baseline: number analyzed (Participants) | 298
  Baseline | 123.5 (115.0)
  4 weeks: number analyzed (Participants) | 163
  4 weeks | 128.8 (95.4)
  8 weeks: number analyzed (Participants) | 178
  8 weeks | 118.6 (90.1)
  24 weeks: number analyzed (Participants) | 188
  24 weeks | 117.9 (70.6)
  52 weeks: number analyzed (Participants) | 142
  52 weeks | 126.5 (103.5)

11. Secondary Outcome: Nutrition Endpoints - Haemoglobin
Description: as for outcome 4
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, and 52 weeks
Population: Among patients in the safety analysis set, 547 patients were included in the efficacy analysis set, excluding 6 patients who were excluded from the efficacy analysis set (Reasons: Unassessable: 5 patients; and off-label use: 1 patient). Among patients in the 547 patients, the patients for which data were obtained at each time frame were analyzed (Baseline:465 patients, 4 weeks:331 patients, 8 weeks:333 patients, 24 weeks:328 patients, 52weeks: 246 patients).
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
g/dL
  Baseline: number analyzed (Participants) | 465
  Baseline | 12.18 (1.99)
  4 weeks: number analyzed (Participants) | 331
  4 weeks | 12.03 (1.84)
  8 weeks: number analyzed (Participants) | 333
  8 weeks | 12.12 (1.95)
  24 weeks: number analyzed (Participants) | 328
  24 weeks | 12.40 (1.96)
  52 weeks: number analyzed (Participants) | 246
  52 weeks | 12.58 (1.88)

12. Secondary Outcome: Patient's Quality of Life - Mental Health (Summary)
Description: Baseline, 8 and 24 weeks after the start of treatment, and at the end of the observation period, the patient was asked to fill out the standard SF-8™ (1 month) to assess the patient's QOL, which was recorded in the survey form for this survey. SF-8™:The Medical Outcomes Study 8-Item Short-Form Health Survey (Japanese version). Items are as follows.
  Physical health (summary):PCS8, Mental health (summary):MCS8, General health:SF8GH, Physical functioning:SF8PF, Role physical:SF8RP, Body pain:SF8BP, Vitality:SF8VT, Social functioning:SF8SF, Mental health:SF8MH, Role emotional:SF8RE.
  MCS8 score is calculated by the following formula (All summed). MCS8 score = (-0.02020×SF8GH)+(-0.19972×SF8PF)+(-0.16579×SF8RP)+(-0.15992×SF8BP)+(0.16737×SF8VT)+(0.27264×SF8SF)+(0.57583×SF8MH)+(0.42927×SF8RE)+4.34744
  The minimum value of MCS8 is 10.108, and the maximum value is 74.511. Higher scores mean a better outcome.
  The means ± SD was calculated by summing the values at each time point.
Time Frame: Baseline, 8 weeks, 24 weeks, and 52 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
score on a scale
  Baseline: number analyzed (Participants) | 517
  Baseline | 44.619 (8.405)
  8 weeks: number analyzed (Participants) | 366
  8 weeks | 47.864 (7.255)
  24 weeks: number analyzed (Participants) | 350
  24 weeks | 49.288 (6.230)
  52 weeks: number analyzed (Participants) | 249
  52 weeks | 49.894 (6.308)

13. Secondary Outcome: Patient's Quality of Life - General Health
Description: Baseline, 8 and 24 weeks after the start of treatment, and at the end of the observation period, the patient was asked to fill out the standard SF-8™ (1 month) to assess the patient's QOL, which was recorded in the survey form for this survey. SF-8™:The Medical Outcomes Study 8-Item Short-Form Health Survey (Japanese version). Items are as follows.
  Physical health (summary):PCS8, Mental health (summary):MCS8, General health:SF8GH, Physical functioning:SF8PF, Role physical:SF8RP, Body pain:SF8BP, Vitality:SF8VT, Social functioning:SF8SF, Mental health:SF8MH, Role emotional:SF8RE.
  SF8GH scores; 1:63.38, 2:58.54, 3:50.27, 4:40.40, 5:34.38, 6:26.89 The minimum value of SF8GH is 26.89, and the maximum value is 63.38. Higher scores mean a better outcome.
  The means ± SD was calculated by summing the values at each time point.
Time Frame: Baseline, 8 weeks, 24 weeks, and 52 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
score on a scale
  Baseline: number analyzed (Participants) | 517
  Baseline | 43.673 (8.513)
  8 weeks: number analyzed (Participants) | 366
  8 weeks | 48.238 (7.395)
  24 weeks: number analyzed (Participants) | 350
  24 weeks | 50.250 (7.306)
  52 weeks: number analyzed (Participants) | 249
  52 weeks | 51.479 (7.030)

14. Secondary Outcome: Patient's Quality of Life - Physical Functioning
Description: Baseline, 8 and 24 weeks after the start of treatment, and at the end of the observation period, the patient was asked to fill out the standard SF-8™ (1 month) to assess the patient's QOL, which was recorded in the survey form for this survey. SF-8™:The Medical Outcomes Study 8-Item Short-Form Health Survey (Japanese version). Items are as follows.
  Physical health (summary):PCS8, Mental health (summary):MCS8, General health:SF8GH, Physical functioning:SF8PF, Role physical:SF8RP, Body pain:SF8BP, Vitality:SF8VT, Social functioning:SF8SF, Mental health:SF8MH, Role emotional:SF8RE.
  SF8PF scores; 1:53.54, 2:47.77, 3:41.45, 4:27.59, 5:16.69 The minimum value of SF8PF is 16.69, and the maximum value is 53.54. Higher scores mean a better outcome.
  The means ± SD was calculated by summing the values at each time point.
Time Frame: Baseline, 8 weeks, 24 weeks, and 52 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
score on a scale
  Baseline: number analyzed (Participants) | 517
  Baseline | 41.941 (10.463)
  8 weeks: number analyzed (Participants) | 366
  8 weeks | 45.630 (8.628)
  24 weeks: number analyzed (Participants) | 350
  24 weeks | 47.438 (7.617)
  52 weeks: number analyzed (Participants) | 249
  52 weeks | 48.325 (7.166)

15. Secondary Outcome: Patient's Quality of Life - Role Physical
Description: Baseline, 8 and 24 weeks after the start of treatment, and at the end of the observation period, the patient was asked to fill out the standard SF-8™ (1 month) to assess the patient's QOL, which was recorded in the survey form for this survey. SF-8™:The Medical Outcomes Study 8-Item Short-Form Health Survey (Japanese version). Items are as follows.
  Physical health (summary):PCS8, Mental health (summary):MCS8, General health:SF8GH, Physical functioning:SF8PF, Role physical:SF8RP, Body pain:SF8BP, Vitality:SF8VT, Social functioning:SF8SF, Mental health:SF8MH, Role emotional:SF8RE.
  SF8RP scores; 1:54.09, 2:47.42, 3:40.65, 4:27.91, 5:21.80. The minimum value of SF8RP is 21.80, and the maximum value is 54.09. Higher scores mean a better outcome.
  The means ± SD was calculated by summing the values at each time point.
Time Frame: Baseline, 8 weeks, 24 weeks, and 52 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
score on a scale
  Baseline: number analyzed (Participants) | 517
  Baseline | 41.325 (10.707)
  8 weeks: number analyzed (Participants) | 366
  8 weeks | 45.253 (8.983)
  24 weeks: number analyzed (Participants) | 350
  24 weeks | 47.371 (8.034)
  52 weeks: number analyzed (Participants) | 249
  52 weeks | 48.222 (7.553)

16. Secondary Outcome: Patient's Quality of Life - Body Pain
Description: Baseline, 8 and 24 weeks after the start of treatment, and at the end of the observation period, the patient was asked to fill out the standard SF-8™ (1 month) to assess the patient's QOL, which was recorded in the survey form for this survey. SF-8™:The Medical Outcomes Study 8-Item Short-Form Health Survey (Japanese version). Items are as follows.
  Physical health (summary):PCS8, Mental health (summary):MCS8, General health:SF8GH, Physical functioning:SF8PF, Role physical:SF8RP, Body pain:SF8BP, Vitality:SF8VT, Social functioning:SF8SF, Mental health:SF8MH, Role emotional:SF8RE.
  SF8BP scores; 1:60.35, 2:52.46, 3:46.10, 4:38.21, 5:31.59, 6:21.68. The minimum value of SF8BP is 21.68, and the maximum value is 60.35. Higher scores mean a better outcome.
  The means ± SD was calculated by summing the values at each time point.
Time Frame: Baseline, 8 weeks, 24 weeks, and 52 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
score on a scale
  Baseline: number analyzed (Participants) | 517
  Baseline | 48.282 (10.178)
  8 weeks: number analyzed (Participants) | 366
  8 weeks | 52.407 (8.162)
  24 weeks: number analyzed (Participants) | 350
  24 weeks | 53.746 (7.906)
  52 weeks: number analyzed (Participants) | 249
  52 weeks | 54.594 (7.852)

17. Secondary Outcome: Patient's Quality of Life - Vitality
Description: Baseline, 8 and 24 weeks after the start of treatment, and at the end of the observation period, the patient was asked to fill out the standard SF-8™ (1 month) to assess the patient's QOL, which was recorded in the survey form for this survey. SF-8™:The Medical Outcomes Study 8-Item Short-Form Health Survey (Japanese version). Items are as follows.
  Physical health (summary):PCS8, Mental health (summary):MCS8, General health:SF8GH, Physical functioning:SF8PF, Role physical:SF8RP, Body pain:SF8BP, Vitality:SF8VT, Social functioning:SF8SF, Mental health:SF8MH, Role emotional:SF8RE.
  SF8VT scores; 1:60.01, 2:53.74, 3:44.48, 4:38.51, 5:28.68. The minimum value of SF8VT is 28.68, and the maximum value is 60.01. Higher scores mean a better outcome.
  The means ± SD was calculated by summing the values at each time point.
Time Frame: Baseline, 8 weeks, 24 weeks, and 52 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
score on a scale
  Baseline: number analyzed (Participants) | 517
  Baseline | 44.425 (8.216)
  8 weeks: number analyzed (Participants) | 366
  8 weeks | 48.408 (7.718)
  24 weeks: number analyzed (Participants) | 350
  24 weeks | 50.263 (7.183)
  52 weeks: number analyzed (Participants) | 249
  52 weeks | 51.463 (6.919)

18. Secondary Outcome: Patient's Quality of Life - Social Functioning
Description: Baseline, 8 and 24 weeks after the start of treatment, and at the end of the observation period, the patient was asked to fill out the standard SF-8™ (1 month) to assess the patient's QOL, which was recorded in the survey form for this survey. SF-8™:The Medical Outcomes Study 8-Item Short-Form Health Survey (Japanese version). Items are as follows.
  Physical health (summary):PCS8, Mental health (summary):MCS8, General health:SF8GH, Physical functioning:SF8PF, Role physical:SF8RP, Body pain:SF8BP, Vitality:SF8VT, Social functioning:SF8SF, Mental health:SF8MH, Role emotional:SF8RE.
  SF8SF scores; 1:55.14, 2:45.60, 3:37.65, 4:29.15, 5:26.00. The minimum value of SF8SF is 26.00, and the maximum value is 55.14. Higher scores mean a better outcome.
  The means ± SD was calculated by summing the values at each time point.
Time Frame: Baseline, 8 weeks, 24 weeks, and 52 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
score on a scale
  Baseline: number analyzed (Participants) | 517
  Baseline | 42.345 (10.332)
  8 weeks: number analyzed (Participants) | 366
  8 weeks | 46.073 (9.255)
  24 weeks: number analyzed (Participants) | 350
  24 weeks | 47.749 (8.393)
  52 weeks: number analyzed (Participants) | 249
  52 weeks | 48.633 (7.973)

19. Secondary Outcome: Patient's Quality of Life - Mental Health
Description: Baseline, 8 and 24 weeks after the start of treatment, and at the end of the observation period, the patient was asked to fill out the standard SF-8™ (1 month) to assess the patient's QOL, which was recorded in the survey form for this survey. SF-8™:The Medical Outcomes Study 8-Item Short-Form Health Survey (Japanese version). Items are as follows.
  Physical health (summary):PCS8, Mental health (summary):MCS8, General health:SF8GH, Physical functioning:SF8PF, Role physical:SF8RP, Body pain:SF8BP, Vitality:SF8VT, Social functioning:SF8SF, Mental health:SF8MH, Role emotional:SF8RE.
  SF8MH scores; 1:56.93, 2:50.72, 3:44.94, 4:36.30, 5:27.59. The minimum value of SF8MH is 27.59, and the maximum value is 56.93. Higher scores mean a better outcome.
  The means ± SD was calculated by summing the values at each time point.
Time Frame: Baseline, 8 weeks, 24 weeks, and 52 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
score on a scale
  Baseline: number analyzed (Participants) | 517
  Baseline | 46.066 (8.459)
  8 weeks: number analyzed (Participants) | 366
  8 weeks | 49.619 (7.245)
  24 weeks: number analyzed (Participants) | 350
  24 weeks | 51.326 (6.267)
  52 weeks: number analyzed (Participants) | 249
  52 weeks | 51.745 (6.395)

20. Secondary Outcome: Patient's Quality of Life - Role Emotional
Description: Baseline, 8 and 24 weeks after the start of treatment, and at the end of the observation period, the patient was asked to fill out the standard SF-8™ (1 month) to assess the patient's QOL, which was recorded in the survey form for this survey. SF-8™:The Medical Outcomes Study 8-Item Short-Form Health Survey (Japanese version). Items are as follows.
  Physical health (summary):PCS8, Mental health (summary):MCS8, General health:SF8GH, Physical functioning:SF8PF, Role physical:SF8RP, Body pain:SF8BP, Vitality:SF8VT, Social functioning:SF8SF, Mental health:SF8MH, Role emotional:SF8RE.
  SF8RE scores; 1:54.19, 2:48.04, 3:42.24, 4:31.42, 5:19.98. The minimum value of SF8RE is 19.98, and the maximum value is 54.19. Higher scores mean a better outcome.
  The means ± SD was calculated by summing the values at each time point.
Time Frame: Baseline, 8 weeks, 24 weeks, and 52 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
score on a scale
  Baseline: number analyzed (Participants) | 517
  Baseline | 43.320 (9.704)
  8 weeks: number analyzed (Participants) | 366
  8 weeks | 47.179 (7.930)
  24 weeks: number analyzed (Participants) | 350
  24 weeks | 48.670 (6.778)
  52 weeks: number analyzed (Participants) | 249
  52 weeks | 49.607 (6.561)

21. Secondary Outcome: Symptoms Related to Exocrine Pancreatic Insufficiency - Frequency of Bowel Movements
Description: as for outcome 9
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, and 52 weeks
Population: Among patients in the safety analysis set, 547 patients were included in the efficacy analysis set, excluding 6 patients who were excluded from the efficacy analysis set (Reasons: Unassessable: 5 patients; and off-label use: 1 patient). Among patients in the 547 patients, the patients for which data were obtained at each time frame were analyzed (Baseline:437 patients, 4 weeks:334 patients, 8 weeks:324 patients, 24 weeks:317 patients, 52weeks: 248 patients).
Measure: Mean (Standard Deviation); unit: times/day
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
times/day
  Baseline: number analyzed (Participants) | 437
  Baseline | 2.37 (1.87)
  4 weeks: number analyzed (Participants) | 334
  4 weeks | 1.82 (1.33)
  8 weeks: number analyzed (Participants) | 324
  8 weeks | 1.77 (1.42)
  24 weeks: number analyzed (Participants) | 317
  24 weeks | 1.51 (0.96)
  52 weeks: number analyzed (Participants) | 248
  52 weeks | 1.43 (0.81)

22. Secondary Outcome: Symptoms Related to Exocrine Pancreatic Insufficiency - Diarrhoea
Description: as for outcome 9
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, and 52 weeks
Population: Among patients in the safety analysis set, 547 patients were included in the efficacy analysis set, excluding 6 patients who were excluded from the efficacy analysis set (Reasons: Unassessable: 5 patients; and off-label use: 1 patient). Among patients in the 547 patients, the patients for which data were obtained at each time frame were analyzed (Baseline:483 patients, 4 weeks:376 patients, 8 weeks:365 patients, 24 weeks:358 patients, 52weeks: 285 patients).
Measure: Number; unit: participants
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
participants
  Baseline, Yes: number analyzed (Participants) | 483
  Baseline, Yes | 187
  Baseline, No: number analyzed (Participants) | 483
  Baseline, No | 296
  4 weeks, Yes: number analyzed (Participants) | 376
  4 weeks, Yes | 81
  4 weeks, No: number analyzed (Participants) | 376
  4 weeks, No | 295
  8 weeks, Yes: number analyzed (Participants) | 365
  8 weeks, Yes | 72
  8 weeks, No: number analyzed (Participants) | 365
  8 weeks, No | 293
  24 weeks, Yes: number analyzed (Participants) | 358
  24 weeks, Yes | 45
  24 weeks, No: number analyzed (Participants) | 358
  24 weeks, No | 313
  52 weeks, Yes: number analyzed (Participants) | 285
  52 weeks, Yes | 29
  52 weeks, No: number analyzed (Participants) | 285
  52 weeks, No | 256

23. Secondary Outcome: Symptoms Related to Exocrine Pancreatic Insufficiency - Foul Stool Odour
Description: as for outcome 9
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, and 52 weeks
Population: Among patients in the safety analysis set, 547 patients were included in the efficacy analysis set, excluding 6 patients who were excluded from the efficacy analysis set (Reasons: Unassessable: 5 patients; and off-label use: 1 patient). Among patients in the 547 patients, the patients for which data were obtained at each time frame were analyzed (Baseline:460 patients, 4 weeks:360 patients, 8 weeks:350 patients, 24 weeks:344 patients, 52weeks: 274 patients).
Measure: Number; unit: participants
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
participants
  Baseline, Yes: number analyzed (Participants) | 460
  Baseline, Yes | 83
  Baseline, No: number analyzed (Participants) | 460
  Baseline, No | 377
  4 weeks, Yes: number analyzed (Participants) | 360
  4 weeks, Yes | 37
  4 weeks, No: number analyzed (Participants) | 360
  4 weeks, No | 323
  8 weeks, Yes: number analyzed (Participants) | 350
  8 weeks, Yes | 30
  8 weeks, No: number analyzed (Participants) | 350
  8 weeks, No | 320
  24 weeks, Yes: number analyzed (Participants) | 344
  24 weeks, Yes | 21
  24 weeks, No: number analyzed (Participants) | 344
  24 weeks, No | 323
  52 weeks, Yes: number analyzed (Participants) | 274
  52 weeks, Yes | 18
  52 weeks, No: number analyzed (Participants) | 274
  52 weeks, No | 256

24. Secondary Outcome: Symptoms Related to Exocrine Pancreatic Insufficiency - Decreased Appetite
Description: as for outcome 9
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, and 52 weeks
Population: Among patients in the safety analysis set, 547 patients were included in the efficacy analysis set, excluding 6 patients who were excluded from the efficacy analysis set (Reasons: Unassessable: 5 patients; and off-label use: 1 patient). Among patients in the 547 patients, the patients for which data were obtained at each time frame were analyzed (Baseline:482 patients, 4 weeks:376 patients, 8 weeks:362 patients, 24 weeks:355 patients, 52weeks: 283 patients).
Measure: Number; unit: participants
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
participants
  Baseline, Yes: number analyzed (Participants) | 482
  Baseline, Yes | 169
  Baseline, No: number analyzed (Participants) | 482
  Baseline, No | 313
  4 weeks, Yes: number analyzed (Participants) | 376
  4 weeks, Yes | 72
  4 weeks, No: number analyzed (Participants) | 376
  4 weeks, No | 304
  8 weeks, Yes: number analyzed (Participants) | 362
  8 weeks, Yes | 58
  8 weeks, No: number analyzed (Participants) | 362
  8 weeks, No | 304
  24 weeks, Yes: number analyzed (Participants) | 355
  24 weeks, Yes | 37
  24 weeks, No: number analyzed (Participants) | 355
  24 weeks, No | 318
  52 weeks, Yes: number analyzed (Participants) | 283
  52 weeks, Yes | 17
  52 weeks, No: number analyzed (Participants) | 283
  52 weeks, No | 266

25. Secondary Outcome: Symptoms Related to Exocrine Pancreatic Insufficiency - Abdominal Distension
Description: as for outcome 9
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, and 52 weeks
Population: Among patients in the safety analysis set, 547 patients were included in the efficacy analysis set, excluding 6 patients who were excluded from the efficacy analysis set (Reasons: Unassessable: 5 patients; and off-label use: 1 patient). Among patients in the 547 patients, the patients for which data were obtained at each time frame were analyzed (Baseline:475 patients, 4 weeks:372 patients, 8 weeks:359 patients, 24 weeks:351 patients, 52weeks: 280 patients).
Measure: Number; unit: participants
Arm/Group | Lipacreon
Number analyzed (Participants) | 547
participants
  Baseline, Yes: number analyzed (Participants) | 475
  Baseline, Yes | 130
  Baseline, No: number analyzed (Participants) | 475
  Baseline, No | 345
  4 weeks, Yes: number analyzed (Participants) | 372
  4 weeks, Yes | 42
  4 weeks, No: number analyzed (Participants) | 372
  4 weeks, No | 330
  8 weeks, Yes: number analyzed (Participants) | 359
  8 weeks, Yes | 37
  8 weeks, No: number analyzed (Participants) | 359
  8 weeks, No | 322
  24 weeks, Yes: number analyzed (Participants) | 351
  24 weeks, Yes | 27
  24 weeks, No: number analyzed (Participants) | 351
  24 weeks, No | 324
  52 weeks, Yes: number analyzed (Participants) | 280
  52 weeks, Yes | 12
  52 weeks, No: number analyzed (Participants) | 280
  52 weeks, No | 268

ADVERSE EVENTS:
Time Frame: From the start of Lipacreon treatment to the end of the observation period or discontinuation. Approximately 52 weeks in the study completers (From date of dosage start, up to 52 weeks).
Arm/Group | LipaCreon
All-Cause Mortality (participants affected / at risk) | 0/553
Serious Adverse Events (participants affected / at risk) | 81/553
Other Adverse Events (participants affected / at risk) | 0/553
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LipaCreon (N=553)
Endocarditis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Bile duct cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 (17)
Pancreatic carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6)
Cerebral infarction (Nervous system disorders) | 2 (2)
Hypogeusia (Nervous system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Mesenteric artery embolism (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 2 (3)
Small intestine ulcer (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1)
Pancreatic duct stenosis (Gastrointestinal disorders) | 1 (1)
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (2)
Cholangitis (Hepatobiliary disorders) | 3 (5)
Cholangitis acute (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 2 (2)
Jaundice cholestatic (Hepatobiliary disorders) | 3 (3)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Skin and subcutaneous tissue disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 2 (2)
Blood albumin decreased (Investigations) | 2 (2)
Low density lipoprotein increased (Investigations) | 1 (1)
Protein total decreased (Investigations) | 3 (3)
Weight decreased (Investigations) | 3 (3)
Weight increased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Chemical peritonitis (Injury, poisoning and procedural complications) | 1 (1)
Activities of daily living impaired (Social circumstances) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No